CLINICAL TRIAL: NCT05286203
Title: Ocular Pathogen and Transcriptome Investigation Using Comprehensive Sequencing
Acronym: OPTICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Nebraska (Other); University of Utah (Other); University of California, Davis (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P0555674
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Uveitis; Infectious Disease
Keywords: Uveitis; Metagenomic deep sequencing; Intraocular infection; MDS
MeSH Terms: conditions — Uveitis; Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Patients enrolled in the trial and randomized to the standard of care (SOC) arm will undergo standard of care testing.
  Interventions: Diagnostic Test: Standard of Care (SOC)
- MDS (Experimental): Patients enrolled in the trial and randomized to the MDS arm will undergo standard of care testing and MDS testing.
  Interventions: Device: Metagenomic Deep Sequencing (MDS)

INTERVENTIONS:
Device: Metagenomic Deep Sequencing (MDS) — MDS is an RNA-seq based testing of ocular fluid or tissue to identify potential infectious pathogens including bacteria, fungi, parasites, and DNA and RNA viruses.
  Arms: MDS
Diagnostic Test: Standard of Care (SOC) — SOC includes any available diagnostic tests, such as Gram stain, cultures, PCRs, that are considered the appropriate testing based on the clinical findings.
  Arms: Standard of Care

SUMMARY:
This is a multi-center randomized controlled evaluator-masked trial designed to compare metagenomic deep sequencing (MDS) versus standard of care testing for improvement of outcomes for intraocular infections. Patients with presumed intraocular infections who meet the eligibility criteria will be randomized to receive MDS testing results or not to receive MDS testing results. All patients will receive standard-of-care testing to guide management. Enrolled patients will be followed at week 2, week 3-6 (randomization visit), and at 4 weeks after the randomization visit. The proportions of patients who received the appropriate therapy and the proportions of patients with improved outcome will be compared between arms. Patient quality of life, MDS performance, and the provider certainly of belief will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Presumed infectious anterior uveitis, or intermediate uveitis, or posterior uveitis, or panuveitis
* Presumed post-operative endophthalmitis
* Unilateral or bilateral
* 18 years and older

Exclusion Criteria:

* Insufficient specimen for MDS
* Age < 18 years of age
* Pregnancy
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 4-week after randomization
  Dichotomous variable (Y/N) as assessed by a masked evaluator
Appropriate therapy | 4-week after randomization
  Dichotomous variable (Y/N) as determined by an independent expert panel

SECONDARY OUTCOMES:
Provider certainty of belief | 4-week after randomization
  Provider certainty of belief that the patient has an infection (continuous variable from 0 to 100%)
Patient quality of life | 4-week after randomization
  As measured by National Eye Institute Vision Function Questionnaire (min = 0, max = 100; higher means better vision function)
Infection status | 4-week after randomization
  Estimated through latent class analysis that compares MDS with traditional tests for presumed ocular infections. Sensitivity and specificity will be reported as percentage (%)
Provider quality of care | 4-week after randomization
  As measured by the World Health Organization Quality of Life Abbreviated Questionnaire (min = 0, max = 100; higher means better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Doan, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shantha JG, Moussa K, Laovirojjanakul W, Yeh S, Tsui E, Chen JL, Vitale AT, Shakoor A, Larochelle M, Niemeyer K, Mentreddy A, Livnat I, Safo M, Ao W, Choo C, Yan D, Zhong L, Chen C, Da Silva K, Reddy AK, Lee J, Sura A, Crowell EL, Qian Y, Sharon Y, Hinterwirth A, Porco T, Arnold BF, Gonzales J, Acharya NR, Lietman TM, Doan T; OPTICS Study Group. The Effect of Metagenomic Sequencing on Patient Clinical Outcomes for Intraocular Infections: A Multicenter Randomized Controlled Trial. Am J Ophthalmol. 2025 Nov;279:100-109. doi: 10.1016/j.ajo.2025.07.003. Epub 2025 Jul 11. PMID 40653257